CLINICAL TRIAL: NCT00298961
Title: Telepsychiatry: Cost Analysis, Quality of Life, Satisfaction and Effectiveness of Psychiatric Consultation Through Videoconference in a Primary Care Setting
Brief Title: Psychiatric Consultation Through Videoconference in a Primary Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Galil Center for Telemedicine and Medical Informatics (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TelepsychiatryCTIL
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Remote Consultation; Community Psychiatry

INTERVENTIONS:
Device: Videoconference equipment FALCON/IP

SUMMARY:
In our study we will aim to examine the issues of cost analysis, quality of life, clinical efficacy and satisfaction of psychiatric consultations through videoconference in a primary care setting in comparison with in-person psychiatric treatment and primary care only. The main hypotheses of the study are: Satisfaction of the patients will increase, the use of telepsychiatry will reduce the costs for the primary and mental health care centers as well as for the patients, the treatment will be as effective as in-person treatment, the number of patients referred to mental health treatment will be higher than that of the previous year, quality of life will improve and that there will be a stigma reduction of mental illness.

DETAILED DESCRIPTION:
Telepsychiatry, as a method which utilizes videoconferencing as a means for consultation, examination and treatment of patients as a substitute for in-person treatment has been in use now for over 40 years. With telepsychiatry there is an attempt to deal with the issues of providing service to patients who reside at a considerable distance from the mental health facilities or that conversely do not call for mental health services for other diverse reasons such as loss of work days, social stigma, travel expenses and so forth.

In Israel, mental health services are provided to 1.5% of the population whereas the incidence in other developed countries is significantly higher, reaching 3-5%, while the prevalence of mental illness in Israel is similar. One can hypothesize that the above factors such as social stigma, mental health care availability, loss of work days and travel expenses all play a role in this. Consequently, patients may prefer to see their primary care physician as an alternative, and according to reports of the Israeli national health services, 30%-50% of visits to the primary care physician are mental health related. Thanks to the technological advances in telecommunications, especially regarding cost reduction and higher bandwidths, there has been a renewed interest in telepsychiatry. However, the issue of the cost effectiveness of telepsychiatry is still controversial. Out of 380 studies on telepsychiatry published from 1956 to 2002, only 12 dealt with the question of cost effectiveness, and among those the results were equivocal. Another question that has scarcely been studied is that of quality of life within telepsychiatry treatment. Finally, the issue of telepsychiatry that is used as a consultation tool in the aid of the primary physician that occurs physically in his own practice is another novel angle we wish to explore. The advantages embodied in this are potentially many - patient discreteness and confidentiality, decrease in expenses and stigma reduction among others.

In our study we will attempt to address the above issues that have not received the focus of attention in many of the published studies so far - cost analysis and quality of life within the context of telepsychiatry consultation in primary care. Additionally, we will address the issues of clinical efficacy and satisfaction (of the primary care provider as well as that of the patient) from the treatment.

Our study hypotheses are:

1. The satisfaction of the patients will increase during the 12 months of study in the group treated by telepsychiatry in comparison with the control groups.
2. Cost analysis - the use of telepsychiatry will reduce the costs for the primary health care centers and/or for the mental health centers: Travel expenses, a decrease in visitations to the primary health care center, a decrease in hospitalizations in general hospitals and/or psychiatric hospitals, a decrease in the number of ancillary tests and of lost work days.
3. Effectiveness of treatment - the mental and physical well being of the patients will improve or at least not be impaired in the group treated by telepsychiatry as compared to the control groups due to the increased availability of the consultation service.
4. The number of patients referred to mental health treatment will be higher than that of the previous year due to the increased availability of telepsychiatry within the primary care setting.
5. The patients will prefer the telepsychiatry service as compared to a referral to a mental health center.
6. Quality of life will improve or it least not be impaired in the group treated by telepsychiatry as compared to the control groups.
7. Stigma reduction - Visitations to the primary health care center as opposed to the mental health center will lower the possibility of the formation of a social stigma of mental disease.

Comparison Groups:

1. Telepsychiatry treated patients within the primary care setting.
2. In-person treated patients by a psychiatrist at the mental health center.
3. Primary care treated patients without a psychiatry consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by the primary care physician.
* Age 18 and over.
* Speak Hebrew.

Exclusion Criteria:

* Patients that suffer from severe dementia.
* Patients suffering from addiction to drugs or alcohol.
* Patients who are deaf, dumb or blind.
* Patients who have a legal guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-05; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) at 0 months, 6 months and 12 months.

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) at 0 months, 6 months and 12 months.
Hamilton Anxiety Rating Scale (HAM-A) at 0 months, 6 months and 12 months.
Hamilton Depression Rating Scale (HAM-D) at 0 months, 6 months and 12 months.
Global satisfaction questionnaire at 0 months, 6 months and 12 months.
General Health Questionnaire 11 (GHQ11) at 0 months, 6 months and 12 months.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-18) at 0 months, 6 months and 12 months.
Costs: Travel expenses, extra consultations, hospitalizations, Medication, loss of work days, medical visitations, ancillary tests such as ECG, lab tests and others at 0 months, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmud Jabarin, MD, Principal Investigator — Sha'ar Menashe Mental Health Center, Israel; Ilan Modai, MD, MHA, Study Chair — Sha'ar Menashe Mental Health Center, Israel; Ehud Susser, MD, Study Chair — Sha'ar Menashe Mental Health Center, Israel
Locations (1):
- Sha'ar Menashe Mental Health Center Ambulatory Clinic, Hadera, Israel

REFERENCES:
- [Background] Hyler SE, Gangure DP, Batchelder ST. Can telepsychiatry replace in-person psychiatric assessments? A review and meta-analysis of comparison studies. CNS Spectr. 2005 May;10(5):403-13. doi: 10.1017/s109285290002277x. PMID 15858458
- [Background] Frueh BC, Deitsch SE, Santos AB, Gold PB, Johnson MR, Meisler N, Magruder KM, Ballenger JC. Procedural and methodological issues in telepsychiatry research and program development. Psychiatr Serv. 2000 Dec;51(12):1522-7. doi: 10.1176/appi.ps.51.12.1522. PMID 11097648
- [Background] Hilty DM, Luo JS, Morache C, Marcelo DA, Nesbitt TS. Telepsychiatry: an overview for psychiatrists. CNS Drugs. 2002;16(8):527-48. doi: 10.2165/00023210-200216080-00003. PMID 12096934
- [Background] May C, Gask L, Atkinson T, Ellis N, Mair F, Esmail A. Resisting and promoting new technologies in clinical practice: the case of telepsychiatry. Soc Sci Med. 2001 Jun;52(12):1889-901. doi: 10.1016/s0277-9536(00)00305-1. PMID 11352414
- [Background] Monnier J, Knapp RG, Frueh BC. Recent advances in telepsychiatry: an updated review. Psychiatr Serv. 2003 Dec;54(12):1604-9. doi: 10.1176/appi.ps.54.12.1604. PMID 14645799
- [Background] Williams TL, May CR, Esmail A. Limitations of patient satisfaction studies in telehealthcare: a systematic review of the literature. Telemed J E Health. 2001 Winter;7(4):293-316. doi: 10.1089/15305620152814700. PMID 11886667
- [Background] Roine R, Ohinmaa A, Hailey D. Assessing telemedicine: a systematic review of the literature. CMAJ. 2001 Sep 18;165(6):765-71. PMID 11584564
- [Background] Simpson J, Doze S, Urness D, Hailey D, Jacobs P. Telepsychiatry as a routine service--the perspective of the patient. J Telemed Telecare. 2001;7(3):155-60. doi: 10.1258/1357633011936318. PMID 11346475
- [Background] Yoshino A, Shigemura J, Kobayashi Y, Nomura S, Shishikura K, Den R, Wakisaka H, Kamata S, Ashida H. Telepsychiatry: assessment of televideo psychiatric interview reliability with present- and next-generation internet infrastructures. Acta Psychiatr Scand. 2001 Sep;104(3):223-6. doi: 10.1034/j.1600-0447.2001.00236.x. PMID 11531660
- [Background] Dongier M, Tempier R, Lalinec-Michaud M, Meunier D. Telepsychiatry: psychiatric consultation through two-way television. A controlled study. Can J Psychiatry. 1986 Feb;31(1):32-4. doi: 10.1177/070674378603100107. PMID 3512068
- [Background] Cruz M, Krupinski EA, Lopez AM, Weinstein RS. A review of the first five years of the University of Arizona telepsychiatry programme. J Telemed Telecare. 2005;11(5):234-9. doi: 10.1258/1357633054471821. PMID 16035965
- [Background] Hyler SE, Gangure DP. A review of the costs of telepsychiatry. Psychiatr Serv. 2003 Jul;54(7):976-80. doi: 10.1176/appi.ps.54.7.976. PMID 12851433
- [Background] Krupinski EA, Barker G, Lopez AM, Weinstein RS. An analysis of unsuccessful teleconsultations. J Telemed Telecare. 2004;10(1):6-10. doi: 10.1258/135763304322764112. PMID 15006208
- [Background] Hilty DM, Marks SL, Urness D, Yellowlees PM, Nesbitt TS. Clinical and educational telepsychiatry applications: a review. Can J Psychiatry. 2004 Jan;49(1):12-23. doi: 10.1177/070674370404900103. PMID 14763673
- [Background] Kennedy C, Yellowlees P. A community-based approach to evaluation of health outcomes and costs for telepsychiatry in a rural population: preliminary results. J Telemed Telecare. 2000;6 Suppl 1:S155-7. doi: 10.1258/1357633001934492. PMID 10794004